CLINICAL TRIAL: NCT02072395
Title: Treatment of Morbid Obesity With Gastric Plication and Gastric Banding
Brief Title: Gastric Plication and Banding
Acronym: GP and Band
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Bradley Needleman, Associate Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012H0003
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; bariatric surgery; gastric banding; gastric plication
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Band/Plication (Experimental): Treatment -- band/plication
  Interventions: Procedure: Plication

INTERVENTIONS:
Procedure: Plication — Plication of the stomach will be performed in conjunction with placement of a gastric band.

SUMMARY:
The purpose of the study is to assess the efficacy of a hybrid laparoscopic surgical procedure for treatment of morbid obesity, Gastric Plication (G)) and Gastric Banding.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* BMI > or = to 30 and co-morbid conditions or BMI > or = to 40
* Ability to provide informed consent
* Willingness to commit to long-term follow-up

Exclusion Criteria:

* Inability to provide informed consent
* Presence of metabolic or medically correctable cause(s) for obesity, such as untreated hypothyroidism or Prader-Willi
* Contraindications to surgery such as myocardial infarction within last 6 months, end stage renal or liver disease, current infection, or other disease states contraindicative to surgery, in the principal investigator's opinion
* Pregnancy
* Plan to become pregnant within two years post-surgery
* Current addiction to drugs or alcohol
* Previous history of any type of bariatric surgery (de novo group only)
* Hiatal hernia > 3 cm

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Weight loss | Two years
  The primary endpoint is weight loss two years post-surgery.
Complications | 2 years
  Intra and post-operative complications will be tracked.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J Needleman, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Background] Chaudhry UI, Osayi SN, Suzo AJ, Noria SF, Mikami DJ, Needleman BJ. Laparoscopic adjustable gastric banded plication: case-matched study from a single U.S. center. Surg Obes Relat Dis. 2015 Jan-Feb;11(1):119-24. doi: 10.1016/j.soard.2014.05.030. Epub 2014 Jun 4. PMID 25443058